CLINICAL TRIAL: NCT06579950
Title: The Effects of Cool Roofs on Health, Environmental, and Economic Outcomes: a Global Multi-center Cluster-randomized Controlled Trial
Brief Title: Assessing the Effects of Cool Roofs on Indoor Environments and Health
Acronym: REFLECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aditi Bunker (Other)
Collaborators: Sika Services AG (Unknown); SOPREMA (Unknown); Engineered Polymer Solutions (EPS B.V.) (Unknown); Resene (Industry); Pacific Community (Other); Habitat for Humanity (Other); The Tindall Foundation (Other); Rutgers University (Other); Boston University (Other); London School of Hygiene and Tropical Medicine (Other); Heidelberg University (Other); Instituto Tecnológico de Hermosillo (Unknown); University of Ouagadougou, Burkina Faso (Other); Indian Institute of Public Health, India (Other)
Responsible Party: Sponsor-Investigator, Aditi Bunker, Co-Principal Investigator, University of Auckland, New Zealand
Organization: University of Auckland, New Zealand (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3728162; 226745/Z/22/Z (Other Grant/Funding Number: Wellcome Trust UK)
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Resting Heart Rate; Blood Glucose Control; Depression; Heat-related Symptoms; Physician Diagnosed Heat-related Illnesses; Food Insecurity; Diet Quality; Health-related Quality of Life; Indoor Thermal Comfort; Coping Ability; Life Satisfaction; Healthcare Provider Utilization; Hospitalization; Systolic Blood Pressure; Diastolic Blood Pressure; Inner Ear Canal Temperature; Dehydration; Sleep Quality; Cognition; Productivity; Aggression; Indoor Air Temperature; Indoor Relative Humidity; Indoor Heat Index; Household Energy Expenditure
Keywords: Hot Temperature; Humidity; Housing; Heart rate; Cardiovascular; Depression; Mental health; Blood glucose; Diabetes; Cool roof; Heat Stress
MeSH Terms: conditions — Depression; Personal Satisfaction; Dehydration; Sleep Initiation and Maintenance Disorders; Aggression; Psychological Well-Being; Diabetes Mellitus; Heat Stress Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Trial participants will be aware of the intervention to which they have been allocated, and the research fieldworkers will be aware of the intervention allocation. The trial steering committee members and trial statistician will remain blinded until the end of trial period and data collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cool roof (Experimental): Households will receive sunlight reflecting 'cool roof' coating on their roofs.
  Interventions: Other: Cool roof
- No cool roof (No Intervention): No cool roof application. Households will keep their original roofing for the duration of the trial.

INTERVENTIONS:
Other: Cool roof — Cool roofs are a sunlight reflecting roof coating that can reduce indoor temperature. Cool roofs have high solar reflectance (reflecting the ultraviolet and visible wavelengths of sunlight, reducing heat transfer to the surface of a roof) and high thermal emittance (radiating absorbed solar energy).
  Arms: Cool roof

SUMMARY:
Ambient air temperatures in Asian, Latin American, African, and Pacific climate hotspots have broken record highs in 2024, driven by man-made climate change. Solutions are needed to reduce heat exposure in communities. Sunlight-reflecting cool roof coatings passively reduce indoor temperatures and energy use to protect home occupants from extreme heat. Occupants living in poor housing conditions globally - for example in informal settlements, slums, and low-socioeconomic households - are especially vulnerable to increased indoor heat exposure.

Heat exposure can instigate and worsen numerous physical, mental and social health conditions. The worst adverse health effects are being experienced in communities least able to adapt to heat exposure. By reducing indoor temperatures, cool roof use can promote physical, mental and social wellbeing in occupants.

The long-term research goal is to identify viable passive housing adaptation technologies with proven health and environmental benefits to reduce the burden of heat stress in communities affected by heat globally. To meet this goal, the investigators will conduct a cluster-randomized controlled trial to establish the effects of cool roof use on health, indoor environment and economic outcomes in four urban climate hotspots: Ouagadougou, Burkina Faso; Hermosillo, Mexico; Ahmedabad, India; and Niue, Oceania.

DETAILED DESCRIPTION:
Increasing heat exposure from climate change is causing and exacerbating heat-related illnesses in millions worldwide - particularly in low resource settings. June 2024 was the 13th consecutive hottest month on record globally - shattering previous records. Heat exposure can instigate and worsen health conditions including cardiovascular, metabolic, endocrine and respiratory disease, heat-related illnesses, pregnancy complications, and mental health conditions. Adaptation is essential for protecting people from increasing heat exposure. The built environment, especially our homes, are ideal for deploying interventions to reduce heat exposure and accelerate adaptation efforts. However, currently there is a lack of evidence on a global scale - generated through empirical studies - guiding the uptake of interventions to reduce heat stress in low resource settings.

Sunlight-reflecting cool roof coatings passively reduce indoor temperatures and lower energy use, offering protection to home occupants from extreme heat. The investigators aim to conduct a global multi-centre cluster-randomized controlled trial investigating the effects of cool-roof use on health, environmental and economic outcomes in four urban climate hotspots - Ouagadougou, Burkina Faso (sub-Saharan Africa), Ahmedabad, India (Asia), Niue (Oceania), and Hermosillo, Mexico (Latin America). The sites represent hotspots where people experience a triple burden from heat exposure, chronic health issues and vulnerable housing conditions (slums, informal settlements and low socioeconomic housing). They also exhibit diversity in climate profiles, housing typology, level of socioeconomic development, population density and rates of urbanisation.

The trial will quantify whether cool roofs are an effective passive home cooling intervention with beneficial health effects for vulnerable populations in four locations. Findings will inform global policy responses on scaling cool roof implementation to protect people from increasing heat exposure driven by climate change.

ELIGIBILITY:
Inclusion Criteria:

* Permanent household resident.

Exclusion Criteria:

* Roof damage, inaccessible or instability of roof adversely affecting cool roof coating application.
* Participant unable to provide written/verbal informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3200 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Resting heart rate | Eight measurements will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  Resting heart rate in beats per minute measured as the average of three readings in the left arm over one hour using Blip portable automated sphygmomanometers.
Blood glucose control | Two measurements will be taken: one at baseline and one in the last month of three consecutive hottest months.
  Three month average of blood glucose in mmol/mol measured as glycosylated hemoglobin (HbA1c) using capillary blood and the HemoCue® HbA1c 501 System.
Depression | Eight measurements will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  Self-reported presence and frequency of symptoms of depression assessed using aggregate score of the Patient Health Questionnaire 9 (PHQ-9). Minimum score of 0 and a maximum score of 27 with a higher score meaning a worse outcome.

SECONDARY OUTCOMES:
Heat-related symptoms | Eight measurements will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  Self-reported heat-related symptoms in the past month, assessed using a recall questionnaire.
Physician diagnosed heat-related illnesses | Eight measurements will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  Self-reported new diagnosis from a medical practitioner of a heat-related illness in the last month assessed using a recall questionnaire.
Food insecurity | Eight measurements will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  Self-reported experience based measure of individual food security assessed using the Food Insecurity Experience Scale (FIES).
Diet quality | Eight measurements will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  Self-reported individual food group consumption in the previous 24 hours assessed using the Diet Quality Questionnaire (DQQ).
Health-related quality of life | Eight measurements will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  Current self-reported health-related quality of life assessed using the EuroQol EQ-5D-5L quality assessment tool. The minimum and maximum scores for the EuroQol EQ-5D-5L quality assessment tool are -0.59 and 1, respectively. A score of 1 represents the best possible health state, while scores below 0 indicate health states that are considered worse than death.
Indoor thermal comfort | Eight measurements will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  Self-reported household heat, humidity and comfort experience over the last four weeks assessed using a recall questionnaire.
Coping ability | Eight measurements will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  Self-reported coping strategies for high indoor temperatures assessed using a recall questionnaire.
Life satisfaction | Eight measurements will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  Current self-reported life satisfaction assessed using the World Values Survey. Values can range from 1 to 10 with a higher score representing greater life satisfaction.
Healthcare provider utilization | Eight measurements will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  Self-reported healthcare provider utilization in the past four weeks assessed using a recall questionnaire.
Hospitalization | Eight measurements will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  Self-reported overnight hospital stay in the past four weeks assessed using a recall questionnaire.
Systolic Blood Pressure | Eight measurements will be taken: one at baseline and seven over 12 months, covering the three consecutive hottest months and four alternate months.
  Maximum blood pressure (mmHg) during systole measured as the average of three readings in the left arm over one hour using Blip portable automated sphygmomanometers.
Diastolic Blood Pressure | Eight measurements will be taken: one at baseline and seven over 12 months, covering the three consecutive hottest months and four alternate months.
  Minimum blood pressure (mmHg) during diastole measured as the average of three readings in the left arm over one hour using Blip portable automated sphygmomanometers.
Cognition | Eight measurements: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  Accuracy and response time to the four-choice Deary-Liewald Test measured using the CogniFit app-based assessment tool.
Inner Ear Canal Temperature | Eight measurements will be taken: one at baseline and seven over 12 months, covering the three consecutive hottest months and four alternate months.
  Internal body temperature (℃) measured once using Braun digital ear thermometer.
Dehydration | Eight measurements will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  Dehydration as indicated by urine specific gravity ≥1.020 measured as urine specific gravity using Siemens Multistix SG dipstick.
Sleep quality | Eight measurements: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  Self-reported sleep distrubance assessed using the Athens Insomnia Scale (AIS). Values range from 0 to 24 with a higher score indicating a worse outcome.
Aggression | Eight measurements: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  Self-reported personal aggresion assessed using the Buss-Perry Aggression Questionnaire-Ultra Short Form (BPAQ-ML).
Productivity | Eight measurements will be taken: one at baseline and seven over 12 months, covering the three consecutive hottest months and four alternate months.
  Self-reported job absenteeism and presenteeism assessed using the Health and Work Performance Questionnaire Short Form (HPQ-SF).
Indoor air temperature | Measurements at 15 minute intervals for 12 months.
  Indoor air temperature (℃) measured using Hobo MX1101 heat and humidity measurement device.
Indoor relative humidity | Measurements at 15 minute intervals for 12 months.
  Ratio of the amount of water vapor present in the air to the greatest amount possible at the same temperature (%) measured using Hobo MX1101 heat and humidity measurement device.
Indoor heat index | Measurements at 15 minute intervals for 12 months.
  Index that combines air temperature and relative humidity (℃) based on temperature and humidity measurements from the Hobo MX1101 heat and humidity measurement device calculated using the formulae endorsed by the US National Oceanic and Atmospheric Administration.
Household energy expenditure | Eight measurements will be taken: one at baseline and seven over 12 months, covering the three consecutive hottest months and four alternate months.
  Self-reported household energy expenditure assessed using a recall questionnaire from the head of the household.

CONTACTS AND LOCATIONS:
Overall Officials: Collin Tukuitonga, Sir. Dr., Principal Investigator — University of Auckland, New Zealand
Locations (4):
- University Joseph Ki-Zerbo, Ouagadougou, Burkina Faso
- Indian Institute of Public Health Gandhinagar, Ahmedabad, Gandhinagar, India
- Instituto Tecnológico de Hermosillo, Hermosillo, Sanora, Mexico
- Niue, Alofi, Niue

IPD SHARING:
Plan to Share IPD: Yes
Data that can be shared unconditionally underpinning the published research articles will be made available to other researchers at the time of publication, and data will be linked via the article DOI. Data that cannot be unconditionally shared upon publication owing to confidentiality or data protection requirements will be identified as such and a contact email will be provided in relevant publications for data access enquiries by other researchers. Individual names of study participants and identifying factors will be removed prior to data sharing.
  It is expected that demographic data of people at the study sites (family size and composition, basic socioeconomic indicators) may contain personally identifiable information and location data. All such data will be removed prior to storage on online data repositories and therefore will be available to be publicly shared at the time of publication of manuscripts.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: At the time of publication.
URL: http://reflect.org.nz